CLINICAL TRIAL: NCT06375915
Title: Single Arm, Multicenter Phase II Study Investigating the Efficacy and Safety of a Novel Therapeutic Scheme in Patients With Unresectable CholAngiocarcinoma: RadioEmbolization in Combination With CisGem and Durvalumab (MEDI4736)
Brief Title: Precision Medicine in Patients With Unresectable CholAngiocarcinoma: RadioEmbolization and Combined Biological Therapy
Acronym: PM-CARE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Francesco De Cobelli (Other)
Collaborators: Cardarelli Hospital (Other); A.O. Ospedale Papa Giovanni XXIII (Other); AOU Pisana, Pisa, Italy (Unknown)
Responsible Party: Sponsor-Investigator, Francesco De Cobelli, MD, Professor, PI, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM-CARE; PNRR-MAD-2022-12375905 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-03-04; First posted 2024-04-19 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: intrahepatic cholangiocarcinoma; precision medicine; combined treatment; radioembolization (TARE); intrahepatic cholangiocarcinoma (iCC); immunotherapy; immunogenicity
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Yttrium-90; durvalumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tretament arm (Experimental): Single arm treatment
  Interventions: Radiation: radioembolization with Y-90; Drug: Durvalumab; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Radiation: radioembolization with Y-90 — Radioembolization with Y-90 will be performed in nominal day 0
Drug: Durvalumab — Following radioembolization, for 6 cycles -intravenous infusion on day 1 of each cycle
Drug: Cisplatin — Following radioembolization, for 6 cycles -intravenous infusion on day 1 and 8 of each cycle
Drug: Gemcitabine — Following radioembolization, for 6 cycles -intravenous infusion on day 1 and 8 of each cycle

SUMMARY:
Underlying disease mechanisms are fundamental for correct treatment selection and patient management in highly invasive and debilitating non-transmissible diseases. Even though overall disease burden of cancer may have decreased due to a higher degree of awareness, the availability of high-quality healthcare and early diagnosis may become challenging in certain neoplasms. Cholangiocarcinoma is usually diagnosed at advanced stages due to non-specific presentation and is frequently refractory to chemotherapy, causing a massive impact on patients and their families. Surgery is currently the only curative treatment but is available to only approximately 30% of patients. The combination of interventional- and immune-oncology to standard of care creates the perfect substrate for synergistic mechanisms to fight tumor growth; in situ cell death following transarterial embolization(TARE) elicits immune mediated response, inflammatory response and biomarkers of oxidative stress and increases antigen presenting T-cells which an anti-anti progam death ligand (PD-L)1 can bind to; standard of care can then add on with its known effects.The rationale of a combined- locoregional and systemic - treatment lies in the synergistic effects of each of the treatments.

DETAILED DESCRIPTION:
Tumors are highly selective and well defined abnormal cellular proliferations in which microenvironment plays an important role in response to treatment. Intrahepatic Cholangiocarcinoma (iCCA), a tumor derived from the epithelia cells of the bile duct, is particularly invasive and malignant. Personalized treatment options with documented efficacy in patients with iCCA are still not available due to the complex and heterogenous molecular pathogenesis which has not been holistically described. Disease models have limited reproducibility; underlying chronic cholestatic disease, chronic inflammation and risk factors contribute to the complexity and diversity of tumor microenvironment. Although novel systemic therapeutic agents show improvement compared to standard of care chemotherapy, a significant percentage of patients still does not respond to treatment, maybe due to molecular/immunologic features which confer resistance. Local treatment prior to systemic therapy has shown to induce subtle changes in the tumor microenvironment and a systemic immune response: engagement of the immune system may therefore lead to enhanced and long term immunosurveillance and therefore, lasting benefits for cancer patients.

Combined systemic treatment with an anti PD-L1, that binds to the programmed cell death protein 1, and the standard of care (SOC) protein kinase inhibitor sorafenib and gemcitabine (which inhibits DNA synthesis), have been used in clinical trials for other primary liver indications and in patients with biliary tract cancers (TOPAZ trial).

Radioembolization (TARE) combines the embolization properties of microspheres with the radiant effect of Yttrium-90 (Y-90). The locally treated tumor tissue is left in place and releases tumor-associated antigens and danger-associated molecular peptides originating from dead or dying cancer cells which promote the activation of antigen presenting cells and anti-tumor CD8+T cells. The resulting development of a systemic immune response following local treatment may lead to tumor regression at different sites than the one treated locally, leading to the so-called abscopal effect.

Comprehensive evaluations in patients undergoing combined treatment may allow a better understanding of tumor pathophysiology as well as the optimization of combined treatment schemes.

This study will investigate the efficacy, primary endpoint overall response rate according to mRECIST (modified Response Evaluation Criteria in Solid Tumors) , and safety of the association of locoregional radioembolization followed by the combination of standard of care (SOC) chemotherapy with Cisplatin and Gemcitabine and durvalumab in patients with liver predominant unresectable intrahepatic cholangiocarcinoma. The biological profile of patients prior to and following locoregional treatment and the effect of systemic therapy will be characterized in terms of potential biomarkers such as quantitative non-invasive radiological based parameters, tumor tissue profiling and evaluation of biological substrates to help define and stratify patients with higher response and better outcome.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (European Union [EU] Data Privacy Directive) obtained from the patient/legal representative prior to performing any protocol related procedures, including screening evaluations.
* Patients with liver predominant intrahepatic cholangiocarcinoma with intermediate/high rate of early recurrence calculated according to https://k-sahara.shinyapps.io/Veryearlyrecurrence/.
* Patients aged > 18 to ≤ 80 at time of study entry;
* Body weight >30kg
* Suspicion or biopsy confirmed diagnosis of iCC, not previously treated with systemic or surgical therapies, including not previously enrolled in another clinical study with an investigational product;
* Preserved liver function as defined as: Child Pugh Class A; Model for End Stage Liver Disease Score (MELD) <10; Future Liver Remnant (FLR) uptake function ≥2.7%/min/m2 on technetium- 99m mebrofenin hepatobiliary scintigraphy and FLR volume> 30% of total functional liver volume for a normal liver, or > 40% of total functional liver volume if the liver has been damaged by chronic liver disease, cholestasis, steatohepatitis or diabetes;
* No technical contraindications to TARE as confirmed by pre-procedural angiographic and scintigraphy;
* DNA tests for hepatitis B virus (HBV) and RNA tests for hepatitis C virus (HCV) negative at Screening;
* Adequate heart and lung function;
* Eastern Cooperative Oncology Group (ECOG) Performance Score 0 or 1;
* Adequate renal and hepatic function as indicated by: serum creatinine <2x upper limit of normal and estimated glomerular filtration rate (eGFR) ≥30ml/min or 1.73m2; measured creatinine clearance (CL) >40 mL/min or calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976*) or by 24-hour urine collection for determination of creatinine clearance; Alkaline phosphatase (ALP), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 5 times the upper limit of normal (ULN) and total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (this will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician);
* Hemoglobin ≥9 g/dL, platelet count ≥75,000/mm3, absolute neutrophil count (ANC) ≥ 1.0 x 109 /L
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Must have a life expectancy of at least 12 weeks

Exclusion Criteria:

* Cancer classified as a combined or mixed type (HCC hepatocelular carcinoma and ICC) at screening -histopathological examination;
* Child-Pugh class B or more or evidence of severe portal hypertension at screening or at any time up to and including baseline;
* History of major gastrointestinal bleeding that required medical intervention within 30 days prior to screening or baseline;
* Known hypersensitivity to tumor specific chemotherapy agents used during the study;
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients;
* Previous allogeneic bone marrow transplant, kidney or liver transplant, i.e. - history of allogenic organ transplantation;
* Active viral, bacterial or fungal infection, clinically relevant for the assessment of suitability;
* Current history or evidence of neuropsychiatric diseases, including depression, schizophrenia,bipolar disorder, impaired cognitive function, dementia, or suicidal tendency;
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis,etc]). The following are exceptions to this criterion: Patients with vitiligo or alopecia; Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement; Any chronic skin condition that does not require systemic therapy; Patients without active disease in the last 5 years may be included but only after consultation with the study physician; Patients with celiac disease controlled by diet alone;
* History of severe cardiovascular disease such as a previous stroke, coronary artery disease requiring surgery, or unresolved arrhythmias within the past 6 months;
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart);
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent
* History of another primary malignancy except for: malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence; Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis;
* Evidence of any hematological malignancy;
* History of active primary immunodeficiency - Positive for human immunodeficiency virus type 1 or 2 (HIV-1, HIV-2) (serum or RNA) - and / or hepatitis B virus surface antigen (HBsAg) positive and/or active Treponema pallidum infection or Mycoplasma (active tuberculosis infection); Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of anti-HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA;
* Alcohol abuse in the 2 months prior to study or other substance abuse in the 6 months prior to the study;
* Pregnant or breastfeeding women or women planning to become pregnant;
* Known bleeding diathesis or history of abnormal bleeding or any other known coagulation abnormality that may contraindicate future surgery or biopsies;
* Use of systemic immunosuppressants or steroids (prednisone equivalent> 10 mg/day);
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion: Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection); Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent; Steroids as premedication for hypersensitivity reactions;
* Active autoimmune conditions
* Patients weighing <30kg will be excluded from enrolment;
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients;
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of Investigational product (IP). Note: Local surgery of isolated lesions for palliative intent is acceptable.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 90 days after the last dose of IP and up to 90 days after the last dose;
* Presence of Hepatopulmonary shunt >20% at diagnostic angiography/99mTC-MAA.
* Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment;
* Presence of Hepatopulmonary shunt >20% at diagnostic angiography/99mTC-MAA;
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 6 months post TARE
  mRECIST criteria on imaging (modified Response Evaluation Criteria in Solid Tumors criteria)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Median progression free survival | Through study completion, an average of 12 months
  mRECIST criteria
Overall response rate | 3 months post TARE
  mRECIST criteria
Overall response rate | 3 months post TARE
  RECIST 1.1 criteria
Overall response rate | Approximately 6 months post TARE
  mRECIST
Overall response rate | Approximately 6 months post TARE
  RECIST 1.1 criteria
Tumor circulating markers tumor tissue-based markers tumor circulating markers tumor tissue-based markers | At the begining of Cycle 1, 2, 3, 4, 5, 6 (each cycle is 21 days)
  Cytokine profile assay
Tumor circulating markers | At the begining of Cycle 1, 2, 3, 4, 5, 6 (each cycle is 21 days)
  Flow cytometry analysis
Tumor tissue based evaluation | During study conduction, at baseline
  Biopsy - histopathology diagnosis
Tumor tissue-based markers tumor tissue-based markers tumor circulating markers tumor tissue-based markers | During study conduction, at baseline
  Biopsy - gene expression
Tumor tissue-based markers tumor tissue-based markers tumor circulating markers tumor tissue-based markers | During study conduction, prior to the begining of Cycle 1 (each cycle is 21 days)
  Biopsy - gene expression
Tumor tissue-based markers tumor circulating markers tumor tissue-based markers | During study conduction, at baseline
  Biopsy - immune landscape
Tumor tissue-based markers tumor circulating markers tumor tissue-based markers | During study conduction, prior to the begining of Cycle 1 (each cycle is 21 days)
  Biopsy - immune landscape
Tumor tissue-based markers tumor circulating markers tumor tissue-based markers | During study conduction, at baseline
  Biopsy - Immuno histochemistry (IHC)
Tumor tissue-based markers tumor circulating markers tumor tissue-based markers | During study conduction, prior to the beginning of Cycle 1 (each cycle is 21 days)
  Biopsy - Immuno histochemistry (IHC)
Quantitative imaging based biomarkers | Through study completion, an average of 2 years
  Software extracted quantitive parameters
Quantitative biomarkers | Through study completion, an average of 2 years
  Imaging based software extracted radiomic features
Overall Survival (OS) | Through study completion, an average of 2 years (right censored)
  Overall Survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No